CLINICAL TRIAL: NCT05344547
Title: Women With Polycystic Ovary Syndrome Are at High Risk to Cardiac Insults
Brief Title: Women With Polycystic Ovary Syndrome Are at High Risk for Cardiac Insults
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amr Fayez Al-kassas, lecturer of Cardiology, Tanta University
Other Study IDs: 35179/1/22
Record Dates: First submitted 2022-04-16; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCOS Patient
  Interventions: Diagnostic Test: Cardiac risk ratio (CRR)
- Non-PCOS Patient
  Interventions: Diagnostic Test: Cardiac risk ratio (CRR)

INTERVENTIONS:
Diagnostic Test: Cardiac risk ratio (CRR) — Cardiac risk ratio (CRR) was calculated according to Genest et al. (23) as serum total cholesterol (TC) level divided by serum high-density lipoprotein-cholesterol (HDL-c) level and woman with CRR at ≥3.5 was considered at risk of cardiac disease (24).

SUMMARY:
Objectives: Evaluation of the cardiovascular (CV) risk in a sample of CV asymptomatic infertile women with polycystic ovary syndrome (PCOS).

Patients & Methods: 100 infertile PCOS women older than 30 years (PCOS group) and 50 fertile non-PCOS women (Non-PCOS group) underwent gynecological and laboratory diagnosis and then underwent a diagnostic protocol consisting of determination of body mass index (BMI), Homeostasis model assessment of insulin resistance (HOMA-IR) scoring and cardiologic evaluation using echocardiography, estimation of carotid artery intima-media thickness (CIMT), coronary artery calcium (CAC) score using multi-slice non-contrast cardiac CT and cardiac risk ratio (CRR). Study outcomes included the incidence of abnormal cardiac risk parameters and the determination of the best minimally invasive modality to be used as a screening test for these women.

DETAILED DESCRIPTION:
Women attending the infertility clinics at Tanta and Benha University Hospitals were eligible for evaluation for PCOS as a cause of infertility. Gynecological evaluation entails data concerning present and past history of menstrual regularity, previous pregnancy for married women, previous investigations or therapies for PCOS or infertility. PCOS was diagnosed depending on the presence of at least two of the Rotterdam criteria

ELIGIBILITY:
Inclusion Criteria:

Infertile PCOS women older than 30 years and free of exclusion criteria were enrolled in the study as PCOS group. Fifty non-PCOS women of age- and BMI cross-matched to the enrolled PCOS women with regular menstrual cycles or fertile if married were collected as control (Non-PCOS) group. Only women who signed the written informed consent will be enrolled in the study.

Exclusion Criteria:

* Age younger than 30 years old, BMI>35 kg/m2, presence of acute or chronic inflammatory diseases, diabetes mellitus, hyperprolactinemia, thyroid dysfunction, Cushing's syndrome, congenital adrenal hyperplasia, adrenal tumor or ovarian tumor, autoimmune disease, malignancy, central nervous system disease, current or previous use of oral contraceptives within 6 months of enrollment were excluded from the study. Patients had congenital cardiac lesions, manifestations of atherosclerosis or family history of cardiac or cerebrovascular insults, ejection fraction <50%, regional wall motion abnormalities and significant valvular diseases were excluded.

Ages: 30 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Women attending the infertility clinics at Tanta and Benha University Hospitals were eligible for evaluation for the PCOS as a cause of infertility. Gynecological evaluation entails data concerning present and past history of menstrual regularity, previous pregnancy for married women, previous investigations or therapies for PCOS or infertility. PCOS was diagnosed depending on the presence of at least two of the Rotterdam criteria
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-03-21 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Abnormal Cardiac Outcomes | 1 to 3 months
  incidence of abnormal cardiac risk parameters among PCOS women who were apparently cardiac free women

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta university, Tanta, El-Gharbyia, Egypt